CLINICAL TRIAL: NCT07214532
Title: SIgnatera-Guided Initiation of Adjuvant CDK4/6 Inhibitor in Intermediate Risk HR+ HER2- Breast Cancer
Brief Title: Signatera-Guided CDK4/6 Inhibitor Therapy in Breast Cancer
Acronym: SIGNAL-ER 101
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-085-NCP
Record Dates: First submitted 2025-09-24; First posted 2025-10-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms; Carcinoma, Ductal, Breast; Receptors, Estrogen (for ER-positive Requirement)
Keywords: ctDNA; Circulating tumor DNA; Signatera; CDK4/6 inhibitor; Ribociclib; Abemaciclib; Molecular residual disease; MRD; Biomarker-guided therapy; Adjuvant therapy; Hormone receptor positive; HER2 negative; Early breast cancer; Intermediate risk breast cancer; breast cancer; Endocrine therapy; Tumor-informed assay
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast

STUDY DESIGN:
Intervention Model Description: This single-arm study uses circulating tumor DNA (ctDNA) testing to guide individualized treatment decisions. All participants undergo ctDNA surveillance every 3 months, with treatment pathways determined by test results rather than randomization. Participants with positive ctDNA receive CDK4/6 inhibitor therapy plus endocrine therapy, while those with negative results continue endocrine therapy alone with ongoing surveillance. Outcomes are compared to historical controls from the NataLEE trial using a non-inferiority design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ctDNA-Guided Therapy (Experimental): All participants receive circulating tumor DNA (ctDNA) testing using Signatera Genome every 3 months to guide treatment decisions. Participants with positive ctDNA results initiate CDK4/6 inhibitor therapy (ribociclib or abemaciclib) in addition to standard endocrine therapy. Participants with negative ctDNA results continue endocrine therapy alone with ongoing ctDNA surveillance. All participants continue their assigned treatment pathway until disease progression, unacceptable toxicity, or study completion.
  Interventions: Device: ctDNA-Guided Treatment Strategy

INTERVENTIONS:
Device: ctDNA-Guided Treatment Strategy — Circulating tumor DNA testing using Signatera Genome assay is performed every 3 months for up to 4 years to guide timing of CDK4/6 inhibitor initiation. Participants with positive ctDNA results initiate CDK4/6 inhibitor therapy (ribociclib or abemaciclib) plus standard endocrine therapy for a minimum of 2 years. Participants with negative ctDNA results continue endocrine therapy alone with ongoing surveillance. CDK4/6 inhibitor selection and endocrine therapy regimen per the physician's choice following standard-of-care guidelines.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ctDNA-guided initiation of CDK4/6 inhibitor therapy using the Signatera™ Designed on Genome test (referred to as "Signatera Genome") in participants with intermediate-risk HR+/HER2- early-stage breast cancer. Based on ctDNA test results, participants will either start CDK4/6 inhibitor therapy in addition to hormone therapy or continue hormone therapy with ongoing ctDNA surveillance. This study will compare outcomes to historical controls from the NataLEE trial to determine whether ctDNA-guided timing maintains efficacy while reducing unnecessary treatment. Participants will be followed for up to 9 years with regular blood draws, hormone therapy, imaging as needed, and quality-of-life assessments.

DETAILED DESCRIPTION:
Participants with intermediate-risk, early-stage HR+/HER2- breast cancer will be enrolled in a prospective, single-arm, multicenter phase II study. Circulating tumor DNA (ctDNA) surveillance will be performed using the Signater Genome assay, which is customized for each participant from archived tumor and matched normal DNA to detect up to 64 tumor-specific variants in plasma.

Participants who are ctDNA positive at baseline will start CDK4/6 inhibitor therapy along with hormone therapy. Those who are ctDNA negative will continue hormone therapy with ctDNA testing every three months. If ctDNA becomes positive during surveillance, participants will first undergo staging to rule out distant disease before beginning CDK4/6 inhibitor therapy in addition to hormone therapy.

All participants will be followed for up to nine years to assess cancer outcomes. Four-year outcomes will be compared to historical controls from the NataLEE trial to evaluate whether ctDNA-guided timing maintains efficacy while reducing unnecessary treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (ICF) obtained prior to any trial-specific screening procedure.
2. Patient is ≥ 18 years-old at the time of ICF signature.
3. Patient is female with known menopausal status at the time of initiation of adjuvant endocrine therapy (ET), or male.
4. Patient with histologically confirmed unilateral and unifocal primary invasive adenocarcinoma of the breast prior to initiating adjuvant chemotherapy, if indicated, or within 6 months of initiating adjuvant endocrine therapy if chemotherapy is not indicated. Patients who receive neoadjuvant endocrine therapy or chemotherapy are allowed to enroll.
5. Patient has breast cancer that is positive for ER and/or PR according to the local laboratory as determined on the most recently analyzed tissue sample.
6. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test (FISH, CISH, or SISH) or an immunohistochemistry (IHC) status of 0 or 1+. If IHC is 2+, a negative in situ hybridization (ISH) test is required to confirm the HER2-negative status.
7. Patient has available archival tumor tissue from the diagnostic biopsy or surgical specimen, for submission to a central laboratory for Signatera testing (unless Signatera Genome clinical testing has already been performed).
8. Patient after surgical resection where tumor was removed completely (i.e., negative microscopic margins on final pathology) and have Anatomic Stage II that is either:

   * N1 or,
   * If N0, T2 or T3 with G2-3 and/or Ki67≥20% (testing for Ki67 not mandatory), excluding G1.

   Notes:
   1. Patients who received neoadjuvant treatment must meet the criteria for stage, grade, Ki67 in any presurgical staging/sample and/or in the surgical specimen.
   2. Categorization into the AJCC 8th edition Anatomic Stage Groups requires determination of the T, N and M categories. ALND can be omitted.
9. Patient has no contraindication to adjuvant ET and is planned to be treated with ET for 5 years (since enrollment date) or more.
10. Provider and patient must be agreeable to initiate CDK4/6 inhibitors only upon ctDNA detection.
11. Patient may have received up to 6 months of standard adjuvant ET at the time of enrollment and any amount of neoadjuvant endocrine therapy.
12. Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
13. Patient must not have a clinical contraindication to ribociclib or abemaciclib.
14. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
15. Women of childbearing potential (CBP) must have a confirmed negative serum pregnancy test within 14 days prior to enrollment.
16. Women of reproductive potential should be advised of the potential risk of CDK4/6 inhibitors to a fetus, and use effective contraception during CDK 4/6 inhibitor therapy.

Exclusion Criteria:

1. Patient has had prior exposure to a CDK4/6 inhibitor.
2. Patient is concurrently using hormone replacement therapy.
3. Patient with a known contraindication or hypersensitivity to ribociclib or abemaciclib as per the FDA indication label.
4. Patients with a multicentric and/or multifocal and synchronous contralateral breast cancer are ineligible.
5. Patient with distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition) and/or evidence of recurrence after curative surgery.
6. Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 5 years before ICF signature. Note: Patients with prior or concurrent in situ malignancies are eligible provided that adequate curative treatment is completed prior to enrollment.
7. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, liver cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infections, active infection requiring systemic antibacterial therapy, etc.) or limit life expectancy to ≤5 years.
8. Patient participated in another interventional study and received treatment with an investigational product (or used an investigational device) within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2037-11-15 (Estimated); Study Completion 2037-12-30 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival | From the date of surgery up to 9 years
  The primary objective of this study is to to evaluate disease free survival (iDFS) in patients with intermediate risk breast cancer receiving standard endocrine therapy with the addition of CDK4/6 inhibitor therapy upon positive ctDNA test results as compared to historical data of treated patients (NataLEE).

CONTACTS AND LOCATIONS:
Overall Officials: Angel Rodriguez, MD, Study Director — Natera, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SA, Liu MC, Aleshin A. Practical recommendations for using ctDNA in clinical decision making. Nature. 2023 Jul;619(7969):259-268. doi: 10.1038/s41586-023-06225-y. Epub 2023 Jul 12. PMID 37438589
- [Background] Kanjanapan Y, Anderson W, Smith M, Green J, Chalker E, Craft P. Real-World Analysis of Breast Cancer Patients Qualifying for Adjuvant CDK4/6 Inhibitors. Clin Breast Cancer. 2025 Feb;25(2):e159-e169.e2. doi: 10.1016/j.clbc.2024.08.022. Epub 2024 Aug 29. PMID 39294027
- [Background] Magbanua MJM, Brown Swigart L, Ahmed Z, Sayaman RW, Renner D, Kalashnikova E, Hirst GL, Yau C, Wolf DM, Li W, Delson AL, Asare S, Liu MC, Albain K, Chien AJ, Forero-Torres A, Isaacs C, Nanda R, Tripathy D, Rodriguez A, Sethi H, Aleshin A, Rabinowitz M, Perlmutter J, Symmans WF, Yee D, Hylton NM, Esserman LJ, DeMichele AM, Rugo HS, van 't Veer LJ. Clinical significance and biology of circulating tumor DNA in high-risk early-stage HER2-negative breast cancer receiving neoadjuvant chemotherapy. Cancer Cell. 2023 Jun 12;41(6):1091-1102.e4. doi: 10.1016/j.ccell.2023.04.008. Epub 2023 May 4. PMID 37146605
- [Background] Cutts R, Ulrich L, Beaney M, Robert M, Coakley M, Bunce C, Crestani GW, Hrebien S, Kalashnikova E, Wu HT, Dashner S, Sethi H, Aleshin A, Liu M, Ring A, Okines A, Smith IE, Barry P, Turner NC, Garcia-Murillas I. Association of post-operative ctDNA detection with outcomes of patients with early breast cancers. ESMO Open. 2024 Sep;9(9):103687. doi: 10.1016/j.esmoop.2024.103687. Epub 2024 Aug 30. PMID 39216186
- [Background] Natarajan A, Tolaney SM. Is adjuvant ribociclib ready for prime time? Ann Oncol. 2024 Dec;35(12):1200-1201. doi: 10.1016/j.annonc.2024.08.2341. Epub 2024 Sep 4. No abstract available. PMID 39241962
- [Background] Johnston SRD, Harbeck N, Toi M, Martin M, O'Shaughnessy J, Rastogi P. Reply to K. Hashimoto and A. Shimomura. J Clin Oncol. 2021 May 1;39(13):1507-1508. doi: 10.1200/JCO.20.03477. Epub 2021 Feb 25. No abstract available. PMID 33630658
- [Background] Kay C, Martinez-Perez C, Dixon JM, Turnbull AK. The Role of Nodes and Nodal Assessment in Diagnosis, Treatment and Prediction in ER+, Node-Positive Breast Cancer. J Pers Med. 2023 Oct 8;13(10):1476. doi: 10.3390/jpm13101476. PMID 37888087
- [Background] Nelson DR, Brown J, Morikawa A, Method M. Breast cancer-specific mortality in early breast cancer as defined by high-risk clinical and pathologic characteristics. PLoS One. 2022 Feb 25;17(2):e0264637. doi: 10.1371/journal.pone.0264637. eCollection 2022. PMID 35213669
- [Background] Smolarz B, Nowak AZ, Romanowicz H. Breast Cancer-Epidemiology, Classification, Pathogenesis and Treatment (Review of Literature). Cancers (Basel). 2022 May 23;14(10):2569. doi: 10.3390/cancers14102569. PMID 35626173
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- See also: Ribociclib, With Adjuvant Endocrine Therapy for ER-positive Breast Cancer (LEADER) — https://clinicaltrials.gov/study/NCT03285412
- See also: D-gSLATfHRR, Estrogen Receptor Positive, HER-2 Negative Breast Cancer (DARE) (DARE) — https://clinicaltrials.gov/study/NCT04567420